CLINICAL TRIAL: NCT05640349
Title: Evaluation of Bacteremia Epidemiology During the COVID Period in One French University Hospital
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22Infectio02
Record Dates: First submitted 2022-12-02; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Bacteremia; Catheter-Related Infections
MeSH Terms: conditions — Bacteremia; Catheter-Related Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Patients with positive blood culture recorded at the microbiology laboratory of University Hospital of Nice during the Covid-19 Pandemic lockdown (between 23/03/2020 and 24/05/2020).
  Interventions: Biological: Positive blood culture
- Control: Patients with positive blood culture recorded at the microbiology laboratory of University Hospital of Nice between 23/03/2019 and 24/05/2019.
  Interventions: Biological: Positive blood culture

INTERVENTIONS:
Biological: Positive blood culture — Positive blood culture recorded at the microbiology laboratory of University Hospital of Nic

SUMMARY:
The main objective of this retrospective cohort is to evaluate the impact of the first epidemic wave during lockdown on bacteremia epidemiology in one French University Hospital.

ELIGIBILITY:
o Inclusion criteria : Patients with positive blood culture recorded at the microbiology laboratory of University Hospital of Nice Aged 18 years

o Exclusion criteria : Patients with negative blood culture recorded at the microbiology laboratory of University Hospital of Nice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of University Hospital of Nice
Sampling Method: Non-Probability Sample
Enrollment: 4200 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Epidemiology of bacteriemia,catheter-related infection and contamination | Day 0
  Describe and compare the incidence and epidemiology of hospital-diagnosed bacteriemia, catheter-related infection and contamination

SECONDARY OUTCOMES:
Characterization of community bacteremia | Day 0
Determined therapeutic actions | Day 0
  Anticipate the diagnostic and therapeutic actions to be taken for future epidemics

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No